CLINICAL TRIAL: NCT05977816
Title: PROPEL-2 Prophylactic Negative Pressure Wound Therapy (NPWT) in Laparotomy Wounds: a Randomised Controlled Trial Comparing Negative Pressure Wound Therapy to Standard Wound Management in Patients Following Midline Laparotomy
Brief Title: PROPEL-2: Prophylactic Negative Pressure Wound Therapy in Laparotomy Wounds
Acronym: PROPEL-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCSI 22-092
Record Dates: First submitted 2023-02-13; First posted 2023-08-04 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Wound Surgical; Wound Infection; Cosmesis
Keywords: Negative Pressure Wound Therapy; Surgical site Infection; Laparotomy; Post-operative Complications; Abdominal Incision; health economics; POSAS; CoPaQ
MeSH Terms: conditions — Surgical Wound; Wound Infection; Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): The wound is dressed using negative pressure wound therapy.
  Interventions: Device: Negative Pressure Wound Therapy
- Standard Wound dressing (Active Comparator): After the skin is closed, the wound is covered using sterile standard gauze dressing.
  Interventions: Other: Standard wound dressing

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — Application of a negative wound pressure therapy dressing to the wound post laparotomy
  Arms: Negative Pressure Wound Therapy
Other: Standard wound dressing — Application of a standard wound dressing to the wound post laparotomy
  Arms: Standard Wound dressing

SUMMARY:
Post-operative wound issues in abdominal surgery have a significant impact on patient outcomes. This study is taking place to investigate if Negative Pressure Wound Therapy (NPWT) dressings reduces Surgical Site Infections, post surgical complications and improves scar appearance compared to standard dressings.

DETAILED DESCRIPTION:
NPWT dressings are designed to remove and absorb any fluid leaking from the wound. This might reduce surgical site infections, improve wound healing and improve scar appearance compared to using standard dressings.

Data is limited in the application of NPWT dressings to laparotomy incisions in the acute and elective care surgery setting. Surgical site infections can complicate a patient's post-operative course significantly, often necessitating a longer length of stay, antibiotic therapy, intervention for wound collections and impair patient mobility and overall recovery.

In addition to this, laparotomy wound complications can possibly delay adjuvant therapy and also increases healthcare costs both as an inpatient and in the community. Despite significant measures to reduce such complications in the form of wound care bundles, changing of gloves prior to wound closure etc., surgical site complications continue to represent a huge healthcare burden.

The Investigators are conducting this study to determine whether NPWT dressings reduce surgical site infections, improve wound healing and scar appearance. This study will also involve a cost-based analysis and seek information from patients on their quality of life. Results from this study will provide evidence on whether these dressings should be used as standard of care for management of surgical laparotomy wounds.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Patient requires visceral abdominal surgery via a midline laparotomy
* Patients who can complete questionnaires

Exclusion Criteria:

• Patients who are unable to adhere to protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Surgical Site Infection (SSI) | 1 month following surgery
  To compare the rate of surgical site infections within 1 month of the surgical procedure, using Negative Pressure Wound Therapy compared to standard dressings. SSIs will be classified according to Centre for Disease Control (CDC) criteria.
Rate of Surgical Site Infection (SSI) | 3 months following surgery
  To compare the rate of surgical site infections within 3 months of the surgical procedure, using Negative Pressure Wound Therapy compared to standard dressings. SSIs will be classified according to Centre for Disease Control (CDC) criteria.
Rate of Surgical Site Infection (SSI) | 6 months following surgery
  To compare the rate of surgical site infections within 6 months of the surgical procedure, using Negative Pressure Wound Therapy compared to standard dressings. SSIs will be classified according to Centre for Disease Control (CDC) criteria.

SECONDARY OUTCOMES:
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | Baseline
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | 1 month following surgery
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | 3 months following surgery
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | 6 months following surgery
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Scar assessment - using the Patient and Observer Scar Assessment Scale (POSAS) | 1 month following surgery
  The POSAS is made up of two scales: the patient scale and the observer scale; each of the six components is scored numerically on a scale of 1 to 10. The component scores are then added together; the worst scar would receive a score of 60, while the best scar would receive a score of 6
Scar assessment - using the Patient and Observer Scar Assessment Scale (POSAS) | 3 months following surgery
  The POSAS is made up of two scales: the patient scale and the observer scale; each of the six components is scored numerically on a scale of 1 to 10. The component scores are then added together; the worst scar would receive a score of 60, while the best scar would receive a score of 6
Scar assessment - using the Patient and Observer Scar Assessment Scale (POSAS) | 6 months following surgery
  The POSAS is made up of two scales: the patient scale and the observer scale; each of the six components is scored numerically on a scale of 1 to 10. The component scores are then added together; the worst scar would receive a score of 60, while the best scar would receive a score of 6
Health-related out-of- Pocket Costs assessed using the Costs for Patients Questionnaire (CoPaQ) | 1 month
  The CoPaQ measures patient and caregivers out-of-pocket expenses (direct and indirect) associated with a health condition
Health-related out-of- Pocket Costs assessed using the Costs for Patients Questionnaire (CoPaQ) | 3 months
  The CoPaQ measures patient and caregivers out-of-pocket expenses (direct and indirect) associated with a health condition
Health-related out-of- Pocket Costs assessed using the Costs for Patients Questionnaire (CoPaQ) | 6 months
  The CoPaQ measures patient and caregivers out-of-pocket expenses (direct and indirect) associated with a health condition
Health Economics evaluation of resource use and cost effectiveness using Negative Pressure Wound Therapy dressings | 6 months
  Investigating resource use and cost effectiveness of single-use, prophylactic negative pressure wound therapy versus standard dressings for midline laparotomy wounds based on length of hospital stay and costs of dressings
Healthcare incremental cost- utility ratio | 6 months
  The incremental cost-effectiveness ratio at 6 months for NPWT vesus standard dressings for patients undergoing laparotomy.The effectiveness will be expressed as quality adjusted life years (QALYs) in a cost-utility analysis. QALYs are a composite measure of outcomes where utilities for health states (on 0-1 scale, where 0 corresponds to death and 1 to full health) act as qualitative weights to combine quantity and quality of life. The number of QALYs in each group will be assessed with the EuroQol 5 Dimensions questionnaire (EQ5D). The EQ-5D measures health status in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression
Healthcare cost-effectiveness ratio at 6 months | 6 months
  Assessment of the cost-effectiveness ratio at 6 months between NPWT dressings compared to standard dressings. The criteria of effectiveness used will be; Length of hospital stay, requirement for return to theatre, requirement for critical care and number of dressings used

CONTACTS AND LOCATIONS:
Overall Officials: Claire Donohoe, PhD, FRCSI, Principal Investigator — Trinity College Dublin /Royal College of Surgeons
Locations (11):
- Ireland (11):
  - Mayo University Hospital, Castlebar
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - University Hospital Galway, Galway
  - Letterkenny University Hospital, Letterkenny
  - University Hospital Limerick, Limerick
  - Sligo University Hospital, Sligo
  - University hospital Kerry, Tralee
  - University Hospital Waterford, Waterford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davey MG, Donlon NE, Walsh SR, Donohoe CL; PROPEL-2 Trial Collaborators. Prophylactic negative pressure wound therapy (NPWT) in laparotomy wounds (PROPEL-2): protocol for a randomized clinical trial. BJS Open. 2024 Jul 2;8(4):zrae081. doi: 10.1093/bjsopen/zrae081. PMID 39178168